CLINICAL TRIAL: NCT01601847
Title: Wheezing in Black Preterm Infants: Impact of Vitamin D Supplementation Strategy
Acronym: D-Wheeze
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Principal Investigator, Anna Maria Hibbs, Assistant Professor of Pediatrics, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R01HL109293 (NIH); R01HL109293 (NIH)
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Wheezing; Allergy
MeSH Terms: conditions — Respiratory Sounds; Hypersensitivity | interventions — Cholecalciferol; Ergocalciferols; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sustained (Active Comparator): Infants will remain on 400 IU/day of cholecalciferol until 6 months of age adjusted for prematurity, regardless of dietary intake
  Interventions: Drug: Cholecalciferol
- Diet-Limited (Placebo Comparator): Infants will receive placebo once their dietary intake of vitamin D has exceeded 200 IU/day
  Interventions: Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Once the dietary intake of vitamin D has exceeded 200 IU/Day, the infants will receive placebo until they are 6 months of age adjusted for prematurity
  Arms: Diet-Limited
Drug: Cholecalciferol — Infants will receive cholecalciferol 400 IU/day PO until they are 6 months of age adjusted for prematurity
  Other Names: D-Vi-Sol; Vitamin D
  Arms: Sustained

SUMMARY:
The goal of this study is to identify a vitamin D supplementation strategy that best promotes the lung, immune, and overall health of black infants born preterm (28-36 weeks gestational age). This is a high risk population that seems to have unique vitamin D needs, and inappropriate supplementation may promote wheezing or allergy. The results of this study will help form nutritional recommendations for the approximately 100,000 black infants born at 30-36 weeks gestational age in the U.S. every year.

DETAILED DESCRIPTION:
Black infants face the highest rates of prematurity in the U.S. (18%), have high rates of prematurity-associated wheezing illnesses, and tend to have lower vitamin D levels. The goal of this [comparative effectiveness] study is to identify a vit. D supplementation strategy that minimizes recurrent wheezing in infancy. Long recognized as important for bone health, a growing body of evidence suggests that vit. D may play a role in the regulation and development of many organ systems. The D pathway regulates lung inflammation and impacts morphogenesis, structure, and cell growth and survival in bronchial smooth muscle. Vit. D exposure has the potential to skew cytokine expression from a Th1 (less allergic) to a Th2 (more allergic) phenotype. Due to their developmental immaturity, preterm infants may be particularly vulnerable to any positive or negative effects of vit. D supplementation on the lung, airway, and immune system. Our preliminary data, supported by the literature, suggests that overly aggressive vit. D supplementation may inadvertently increase wheezing in infancy in black, but not white, preterm infants; however, vit. D deficiency could theoretically also increase wheezing via vulnerability to respiratory pathogens. The proposed study is a randomized clinical trial comparing the effect of two different enteral vitamin D supplementation strategies on recurrent wheezing in infancy in 300 black infants born preterm at 28 0/7-36 6/7 wks gestational age, a population for whom neither vit. D requirements nor optimal vit. D serum levels have been established. The investigators will test two strategies: (I) sustained supplementation until 6 mo. of age adjusted for prematurity, and (II) cessation of supplementation when a minimum dietary intake of 200 IU/day is reached. The specific aims are to characterize the effect of each strategy on (aim 1) recurrent wheezing and (aim 2) allergic sensitization and atopy. The investigators will (aim 3) explore the relationship between vit. D serum levels and recurrent wheezing. The investigators hypothesize that strategy II will be more effective in promoting pulmonary health by minimizing recurrent wheezing, allergic sensitization, and overall healthcare utilization, and will be sufficient to prevent clinical vit. D deficiency. The investigators also hypothesize that optimal vit. D serum levels will be lower than the norms for other populations.

ELIGIBILITY:
Inclusion criteria:

1. 28 0/7-36 6/7 weeks gestational age (GA) at birth;
2. family identifies the child as black or African American;
3. < 28 days of supplemental oxygen (subsequent oxygen therapy for < 72 hrs for a brief subsequent illness or surgery will be allowed);
4. admitted to a participating site NICU, special care nursery, transitional care nursery, or well-baby nursery as a neonate; and
5. < 40 weeks corrected GA at enrollment.

Exclusion criteria:

1. BPD (> 28 days of supplemental oxygen);
2. pre-existing diagnosis of moderate to severe osteopenia of prematurity and/or alkaline phosphatase > 700;
3. history of fracture;
4. gastrointestinal surgery, including for NEC;
5. known gastrointestinal malabsorption;
6. major congenital anomaly;
7. congenital pulmonary or airway disorder (e.g., cystic fibrosis, tracheomalacia, swallowing disorder, bronchopulmonary sequestration);
8. documented wheezing or stridor prior to enrollment;
9. previous vit. D supplementation with > 400 IU/day;
10. family plans to move more than 60 miles from CWRU or other pre-defined radius at other sites;
11. baseline hypo- or hypercalcemia, hypo- or hyperphosphatemia; and
12. baseline 25(OH) D level < 10 ng/ml.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2013-01; Primary Completion 2017-03-12 (Actual); Study Completion 2017-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Hibbs, MD, MSCE, Principal Investigator — Case Western Reserve University
Locations (5):
- United States (5):
  - Montefiore Medical Center, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - University Hospitals, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Benson AC, Chen Z, Minich NM, Tatsuoka C, Furman L, Ross K, Hibbs AM. Human milk feeding and wheeze in Black infants born preterm. J Perinatol. 2022 Nov;42(11):1480-1484. doi: 10.1038/s41372-022-01471-w. Epub 2022 Aug 4. PMID 35927485
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Ledingham L, Tatsuoka C, Minich N, Ross KR, Kerns LA, Wagner CL, Fuloria M, Groh-Wargo S, Zimmerman T, Hibbs AM. Burden of prematurity-associated recurrent wheezing: caregiver missed work in the D-Wheeze trial. J Perinatol. 2021 Jan;41(1):69-76. doi: 10.1038/s41372-020-0729-7. Epub 2020 Jul 21. PMID 32694857
- [Derived] Hibbs AM, Ross K, Kerns LA, Wagner C, Fuloria M, Groh-Wargo S, Zimmerman T, Minich N, Tatsuoka C. Effect of Vitamin D Supplementation on Recurrent Wheezing in Black Infants Who Were Born Preterm: The D-Wheeze Randomized Clinical Trial. JAMA. 2018 May 22;319(20):2086-2094. doi: 10.1001/jama.2018.5729. PMID 29800180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants were recruited from participating NICUs, special care nurseries, and well-baby nurseries.
Pre-assignment Details: If all eligibility labs were not available from routine clinical care, parents were consented prior to obtaining the remaining eligibility labs. If those post-consent laboratory results made the infant ineligible, they were not randomized.
Groups:
- Sustained: Infants will remain on 400 IU/day of cholecalciferol until 6 months of age adjusted for prematurity, regardless of dietary intake
  Cholecalciferol: Infants will receive cholecalciferol 400 IU/day PO until they are 6 months of age adjusted for prematurity.
  Exclusively breastfed infants receive 400 IU of vitamin D daily as needed beyond 6 months adjusted age for the duration of the study.
- Diet-Limited: Infants will receive placebo once their dietary intake of vitamin D has exceeded 200 IU/day
  Cholecalciferol: Once the dietary intake of vitamin D has exceeded 200 IU/Day from formula or fortifiers, the infants will receive placebo until they are 6 months of age adjusted for prematurity.
  Exclusively breastfed infants receive 400 IU of vitamin D daily as needed beyond 6 months adjusted age for the duration of the study.
Period: Overall Study
Arm/Group | Sustained | Diet-Limited
Started | 153 | 147
Completed | 140 | 137
Not Completed | 13 | 10
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 11 | 7
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: One infant was withdrawn from the study prior to completion of the baseline questionnaire a data collection, and is not included all rows in this table.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sustained | Diet-Limited | Total
Number analyzed (Participants) | 153 | 147 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 153 | 147 | 300
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One infant withdrew before completion of all baseline data forms.
  Participants
    number analyzed (Participants) | 153 | 146 | 299
    Female | 76 | 57 | 133
    Male | 77 | 89 | 166
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 153 | 147 | 300
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Gestational age at birth [Median (Full Range); unit: weeks] | 33.00 [29.14 to 36.86] | 33.50 [28.00 to 36.86] | 33.14 [28.00 to 36.86]
Birth weight [Median (Full Range); unit: kg] — Population: One infant was withdrawn before all baseline/inpatient data capture forms were completed.
  kg
    number analyzed (Participants) | 153 | 146 | 299
    (all) | 1.84 [0.82 to 4.05] | 1.96 [0.79 to 3.62] | 1.87 [0.79 to 4.05]
Multiple birth (twins and triplets) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: One infant withdrew before completion of all baseline data forms.
  Participants
    number analyzed (Participants) | 153 | 146 | 299
    (all) | 58 | 38 | 96
Antenatal steroids [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: One infant withdrew before completion of all baseline data forms.
  Participants
    number analyzed (Participants) | 153 | 146 | 299
    (all) | 82 | 78 | 160
History of ventilator support [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: One infant withdrew before completion of all baseline data forms.
  Participants
    number analyzed (Participants) | 153 | 146 | 299
    (all) | 27 | 26 | 53
History of oxygen administration [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: One infant withdrew before completion of all baseline data forms.
  Participants
    number analyzed (Participants) | 153 | 146 | 299
    (all) | 66 | 53 | 119
Receiving maternal breast milk at randomization [Count of Participants; unit: Participants] | 107 | 104 | 211
Discharge season (Oct-March) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: One infant withdrew before completion of all baseline data forms.
  Participants
    number analyzed (Participants) | 153 | 146 | 299
    (all) | 69 | 67 | 136
Calcium (mg/dl) [Median (Full Range); unit: mg/dl] | 9.5 [7.2 to 10.8] | 9.5 [7.1 to 10.7] | 9.5 [7.1 to 10.8]
Phosphorus (mg/dl) [Median (Full Range); unit: mg/dl] | 7.0 [3.5 to 8.9] | 6.9 [3.6 to 8.9] | 7.0 [3.5 to 8.9]
Alkaline phosphatase (U/L) [Median (Full Range); unit: U/L] | 268 [128 to 686] | 257 [70 to 563] | 263 [70 to 686]
Total circulating 25(OH)D (ng/ml) [Median (Full Range); unit: ng/ml] | 19.1 [10.0 to 71.0] | 21.0 [10.0 to 50.0] | 20.2 [10.0 to 71.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Infants With Recurrent Wheezing
Description: Recurrent wheezing was defined as more than 1 episode of wheezing reported during the study period. Separate episodes were defined as occurring at least 2 weeks apart.
Time Frame: up to 12 months adjusted age
Population: Infants that were withdrawn, completely lost to follow-up, who died, or for whom recurrent wheezing status was indeterminate due to a missing 12 month visit (n=8) were not included in the primary analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Sustained | Diet-Limited
Number analyzed (Participants) | 135 | 134
Participants | 42 | 56
Statistical Analysis 1: Comparison: Sustained vs Diet-Limited; Test type: Superiority; p = 0.02, Poisson; Poisson regression using GEE with robust variance estimation (e.g. Zou, American Journal Epidemiology, 2004); Risk Ratio (RR) = 0.66, 95% CI 2-sided [0.47 to 0.94]
Statistical Analysis 2: Comparison: Sustained vs Diet-Limited; Test type: Superiority; p = 0.0185, logistic regression with GEE; Odds Ratio (OR) = 0.522, 95% CI 2-sided [0.304 to 0.897]

2. Secondary Outcome: Number With Infants With Allergic Sensitization as Measured by the PhadiaTop Infant Assay
Description: Measured using the Phadiatop Infant IgE panel
Time Frame: Measured at the 12 month adjusted age visit
Population: Positive result is >0.35 U/L PAU/l
Measure: Count of Participants; unit: Participants
Arm/Group | Sustained | Diet-Limited
Number analyzed (Participants) | 116 | 112
Participants | 7 | 3
Statistical Analysis 1: Comparison: Sustained vs Diet-Limited; For secondary outcomes, GEE is used to assess randomization arm association; Test type: Superiority; p = 0.228, Regression, Logistic

3. Secondary Outcome: Bone Density
Description: Measured by bone speed of sound (ultrasound)
Time Frame: Measured at the 12 month adjusted age visit
Population: Bone density was not performed if (1) infant could not come to the clinic for their 12 month visit and the visit was done in the home (2) they missed their 12 month visit (3) the ultrasound was under repair, or (4) infant could not participate with the ultrasound to get a sufficient quality reading.
Measure: Median (Full Range); unit: m/s
Arm/Group | Sustained | Diet-Limited
Number analyzed (Participants) | 105 | 107
m/s | 3155 [2908 to 3409] | 3149 [2898 to 3351]
Statistical Analysis 1: Comparison: Sustained vs Diet-Limited; Test type: Superiority; p = 0.798, Regression, Logistic

ADVERSE EVENTS:
Time Frame: Up to 12 months adjusted age
Description: Study personnel screened for adverse events at each study visit. Adverse event categories/organ systems are not mutually exclusive (for instance, an AE could be coded under both respiratory and infectious categories). All significant associated symptoms/findings were coded for each (S)AE.
  36 patients in the Sustained arm had a total of 44 SAEs; 38 patients in the Diet-Limited arm had a total of 56 SAEs. Some patients experienced more than one SAE.
Arm/Group | Sustained | Diet-Limited
All-Cause Mortality (participants affected / at risk) | 1/153 | 0/147
Serious Adverse Events (participants affected / at risk) | 36/153 | 38/147
Other Adverse Events (participants affected / at risk) | 123/153 | 123/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sustained (N=153) | Diet-Limited (N=147)
Asthma or Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 13 (21)
Apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Upper Respiratory Infection (Infections and infestations) | 8 (8) | 13 (16)
Lower Respiratory Infection (Infections and infestations) | 11 (11) | 18 (27)
Pulmonary, not otherwise specified (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) — This category was coded if the event did not fit in the other pre-specified pulmonary categories for infections, wheezing, or apnea.
ALTE or BRUE (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4) — "Apparent Life Threatening Event" or "Brief Resolved Unexplained Event." The American Academy of Pediatrics preferred terminology changed during the study.
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea, non-infectious (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting, non-infectious (Gastrointestinal disorders) | 3 (3) | 1 (1)
GI, not otherwise specified (Gastrointestinal disorders) | 7 (7) | 2 (2) — This category was coded if the condition did not fit into the other pre-specified GI categories
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 2 (2)
Hypercalcemia (Endocrine disorders) | 0 (0) | 1 (1)
GI infection (Infections and infestations) | 1 (1) | 0 (0)
Other Infection (Infections and infestations) | 3 (3) | 7 (9) — This category was coded if the infection was not described by other pre-specified infection categories.
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Neurologic, not otherwise specified (Nervous system disorders) | 1 (1) | 1 (1) — This category was coded if the condition was not described by another pre-existing neurologic category.
Fracture (bone) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Failure to Thrive (General disorders) | 4 (7) | 1 (1)
Other (not classified elsewhere) (General disorders) | 6 (6) | 3 (3) — This category was coded if the important signs or symptoms related to the event were was not otherwise described by other pre-existing categories.
Trauma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Vision problem (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sustained (N=153) | Diet-Limited (N=147)
Asthma or Wheezing (Respiratory, thoracic and mediastinal disorders) | 38 (65) | 36 (60)
Upper Respiratory Infection (Infections and infestations) | 84 (163) | 78 (155)
Lower Respiratory Infection (Infections and infestations) | 27 (39) | 23 (31)
Constipation (Gastrointestinal disorders) | 7 (7) | 9 (9)
Diarrhea, non-infectious (Gastrointestinal disorders) | 4 (4) | 16 (16)
Vomiting, non-infectious (Gastrointestinal disorders) | 9 (11) | 19 (21)
GI, not otherwise specified (Gastrointestinal disorders) | 8 (10) | 17 (17) — This category was coded if the event was not described by the other GI categories.
Elevated alkaline phosphatase (Endocrine disorders) | 13 (14) | 12 (14)
Hypercalcemia (Endocrine disorders) | 27 (27) | 25 (29)
GI Infection (Infections and infestations) | 13 (15) | 14 (17)
Infection, not otherwise specified (Infections and infestations) | 44 (63) | 51 (68) — This category was coded if the event was not described by another infection category.
Anemia (Blood and lymphatic system disorders) | 10 (10) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 36 (47) | 42 (56)
Other AE (General disorders) | 19 (22) | 22 (25) — This category was coded if the relevant signs/symptoms of the AE were not otherwise captured by other categories.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT01601847/Prot_SAP_000.pdf